CLINICAL TRIAL: NCT04447560
Title: Effects of Erector Spinae Plane Block on Sympathectomy in Off Pump Coronary Artery Bypass Surgery
Brief Title: Effects of Erector Spinae Plane Block Method Used in Pain Management in Heart Surgery on Vascular Diameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Kamil Darcin, Assistant professor, Koç University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ESPCVS01
Record Dates: First submitted 2020-06-01; First posted 2020-06-25 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease; Erector Spinae Plane Block; Bypass Extremity Graft
Keywords: Cardiac anesthesia; Sympathectomy; Off-pump coroner artery by-pass surgery
MeSH Terms: conditions — Coronary Artery Disease | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: The study is planned as prospective. Aged between 18-75, ASA III risk group and are undergoing off pump coronary artery bypass grafting surgery are selected for the study. Who are allergic to planned-medications, chronic opioid or opioid receptor agonist users, those with preoperative neuropathies, psychiatric diseases will be excluded. Electrocardiography and pulse oximetry monitorization is performed in the recovery room where a peripheric intravenous line is opened afterwards. High frequency (12-24 MHz) linear probe is used for measurements. Images will be recorded by USG from the 3., 4. and 5. intercostal spaces for the LIMA and RIMA and 3cm proximal to the wrist for the right and left radial arteries. After images are saved, the researcher will perform ESP block with USG. ESP block will be performed to right and left sides equally with 40ml %0.25 bupivacaine in total. Artery images will be recorded again by the same researcher after 45 minutes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Erector Spinae Plane Block (Experimental): One researcher will record the artery images as explained in the protocol before and after the plane block and two researchers will measure the radius and area of those vessels separately.
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — One researcher will record the artery images as explained in the protocol and two researchers will measure the radius and area of those vessels separately. Researchers who are measuring the radius and area of vessels won't know whether those images belong to pre or post- ESP block. The results two researchers measure will be compared statistically and if there are no statistically significant differences, the mean value of their separate recordings will be taken into account for the statistical analysis.
  Other Names: Bupivacaine

SUMMARY:
Off-pump coronary artery bypass grafting (OPCABG) is a bypass method performed on the working heart. Pain is a frequently seen side effect experienced following this surgery. Erector spinae plane block is our analgesia method that the investigators routinely perform prior to the surgery to overcome this problem. In this method, analgesic medication is given via a needle in between the two superficial muscle groups (erector spinae muscles) located in participants back. The investigators believe this method not only provides pain relief, but also is beneficial (dilating) on the vessels that will be used for bypassing the clogged vessels during the surgery. The investigators aimed to measure some parameters in this routine procedure before and after performing the analgesic method with an ultrasound (imaging with sound waves).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are aged between 18-75,
* ASA III
* Patients who are undergoing off pump coronary artery bypass grafting surgery

Exclusion Criteria:

* Patients who are allergic to planned-medications,
* those with previous cardiac surgery,
* patients undergoing emergency surgery,
* uncontrolled diabetes mellitus,
* chronic opioid or opioid receptor agonist users,
* those with pre-operative neuropathies, psychiatric diseases,
* non-communicable patients and
* those who refuse to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Effect of erector spinae plane (ESP) block on the change in diameters of mammarian arteries and radial arteries | The first measurement will be done in the pre-operative preparation room for each participant, and block will be performed in sitting position by an experienced anesthesiologist. Second measurement will be done 45 minutes after performing the ESP block
  Linear probe is used for measurements. Images will be recorded by ultrasound from the third, fourth and fifth intercostal spaces for the LIMA and RIMA and 3cm proximal to the wrist for the right and left radial arteries. After images are saved, the researcher will perform ESP block with USG. Linear/convex probe is used to place the needle parasagittally 3 cm lateral to T5 spinous processes. ESP block will be performed to right and left sides equally with 40ml %0.25 bupivacaine in total, to the fascial plane between the transverse process and erector spinae muscle. Artery images will be recorded again by the same researcher after 45 minutes.For the recordings, one researcher will record the images as explained in the protocol and two researchers will measure the records separately. The results measured in millimeters by two researchers will be compared statistically and if there is no significant difference, the average value of the records will be used for statistical analysis.

SECONDARY OUTCOMES:
Measurement of Mean Arterial Pressure on basis, 5,10,15,20,25,30,35,40,45 minutes after the Erector Spinae Plane block | The first measurement will be done in the pre-operative preparation room for each participant, and block will be performed. After the block, a measurement will be made every 5 minutes. The last measurement will be made 45 minutes after the block.
  When each participant comes to the preoperative preparation room, the mean arterial pressure will be measured in mmHg. Then the erector spinae plane block will be performed. After the block is performed, a measurement will be recorded every 5 minutes. The last measurement will be done 45 minutes after the block is performed.
Measurement of Mean Heart Rate on basis, 5,10,15,20,25,30,35,40,45 minutes after the Erector Spinae Plane block. | The first measurement will be done in the pre-operative preparation room for each participant, and block will be performed. After the block, a measurement will be made every 5 minutes. The last measurement will be made 45 minutes after the block.
  When each participant comes to the preoperative preparation room, the heart rate will be measured in per minute. Then the erector spinae plane block will be performed. After the block is performed, a measurement will be recorded every 5 minutes. The last measurement will be done 45 minutes after the block is performed.
Measurement of Pulse Oxymetri on basis, 5,10,15,20,25,30,35,40,45 minutes after the Erector Spinae Plane block. | The first measurement will be done in the pre-operative preparation room for each participant, and block will be performed. After the block, a measurement will be made every 5 minutes. The last measurement will be made 45 minutes after the block.
  When each participant comes to the preoperative preparation room, the pulse oximetry will be measured. Then the erector spinae plane block will be performed. After the block is performed, a measurement will be recorded every 5 minutes. The last measurement will be done 45 minutes after the block is performed.

CONTACTS AND LOCATIONS:
Overall Officials: Ömür Erçelen, Study Director — Koç University
Locations (1):
- Koc University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting from 6 months after publication for 5 years
Access Criteria: No access criteria

REFERENCES:
- [Background] Alvarez J, Hernandez B, Atanassoff PG. High thoracic epidural anesthesia and coronary artery disease in surgical and non-surgical patients. Curr Opin Anaesthesiol. 2005 Oct;18(5):501-6. doi: 10.1097/01.aco.0000183104.73931.22. PMID 16534283
- [Background] Bourke T, Vaseghi M, Michowitz Y, Sankhla V, Shah M, Swapna N, Boyle NG, Mahajan A, Narasimhan C, Lokhandwala Y, Shivkumar K. Neuraxial modulation for refractory ventricular arrhythmias: value of thoracic epidural anesthesia and surgical left cardiac sympathetic denervation. Circulation. 2010 Jun 1;121(21):2255-62. doi: 10.1161/CIRCULATIONAHA.109.929703. Epub 2010 May 17. PMID 20479150
- [Background] Nagaraja PS, Ragavendran S, Singh NG, Asai O, Bhavya G, Manjunath N, Rajesh K. Comparison of continuous thoracic epidural analgesia with bilateral erector spinae plane block for perioperative pain management in cardiac surgery. Ann Card Anaesth. 2018 Jul-Sep;21(3):323-327. doi: 10.4103/aca.ACA_16_18. PMID 30052229
- [Background] Krishna SN, Chauhan S, Bhoi D, Kaushal B, Hasija S, Sangdup T, Bisoi AK. Bilateral Erector Spinae Plane Block for Acute Post-Surgical Pain in Adult Cardiac Surgical Patients: A Randomized Controlled Trial. J Cardiothorac Vasc Anesth. 2019 Feb;33(2):368-375. doi: 10.1053/j.jvca.2018.05.050. Epub 2018 Jun 4. PMID 30055991
- [Background] Smith LM, Barrington MJ; St Vincent's Hospital, Melbourne. Ultrasound-guided blocks for cardiovascular surgery: which block for which patient? Curr Opin Anaesthesiol. 2020 Feb;33(1):64-70. doi: 10.1097/ACO.0000000000000818. PMID 31833864
- [Result] Wink J, Veering BT, Aarts LPHJ, Wouters PF. Effects of Thoracic Epidural Anesthesia on Neuronal Cardiac Regulation and Cardiac Function. Anesthesiology. 2019 Mar;130(3):472-491. doi: 10.1097/ALN.0000000000002558. PMID 30676423

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/60/NCT04447560/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/60/NCT04447560/ICF_001.pdf